CLINICAL TRIAL: NCT04065724
Title: An Exercise Programme for People With Severe Peripheral Neuropathy and Diabetic Foot Ulcers - a Case Series on Feasibility and Safety
Brief Title: Exercise for People With Peripheral Neuropathy and Diabetic Foot Ulcers - a Case Series on Feasibility and Safety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Københavns Kommune (Other)
Collaborators: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Kajsa Lindberg, PT, supervisor, Københavns Kommune
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: KoebenhavnsKommune
Record Dates: First submitted 2019-03-12; First posted 2019-08-22 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Diabetes Mellitus; Foot Ulcer
Keywords: diabetes mellitus; foot ulcer; resistance training; exercise
MeSH Terms: conditions — Diabetes Mellitus; Foot Ulcer; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Physical training resistance and aerobic (Other): Physical training as resistance and aerobic training
  Interventions: Other: Physical training as resistance and aerobic training.

INTERVENTIONS:
Other: Physical training as resistance and aerobic training.

SUMMARY:
Physical training is one of the cornerstones within the treatment of diabetes, as well as medicine and diet modification, and the effect is well documented. Nevertheless people with diabetes with foot ulcers are urged to lessen their level of physical activity, to reduce pressure on footbed and thereby achieve fastest possible healing.

Purpose: The primarily purpose is to investigate the feasibility of implementing safe, progressive resistance training, combined with exercises for ankle mobility and aerobic training, for people with diabetes and foot ulcers, without compromising the ulcer. The secondarily purpose is to investigate whether this form of training is effective on improving muscle strength, as to if limitations in everyday life diminishes.

The hypothesis is, that it is possible to implement a structured exercise program without compromising the diabetic ulcer.

DETAILED DESCRIPTION:
Background:

Physical training is one of the cornerstones within the treatment of diabetes, as well as medicine and diet modification, and the effect is well documented in terms of improved glycemic control, loss of fat tissue, lower content of triglycerides in blood, improved insulin sensitivity, and lower diabetes related mortality. Nevertheless people with diabetes and foot ulcers are urged to lessen their level of physical activity, to reduce pressure and thereby achieve fastest possible healing. Most ulcers occur at the footbed and the rationale is that the pressure on the ulcer area should be minimized to achieve healing.

Purpose: The primarily purpose of the study is to investigate the feasibility of implementing progressive resistance training, combined with exercises for ankle mobility and aerobic training, for people with diabetes and foot ulcers, without compromising the ulcer. The secondarily purpose is to investigate whether this form of training is effective on the following:

* Muscle strength
* Limitations in activity
* Participants´satisfaction The hypothesis is, that it is possible to implement a structured exercise program and achieve improved muscle strength for this population, without compromising the diabetic ulcer.

Material and methods:

* Design:The study is a prospective intervention study. This particular study is the pilot study and has focus on feasibility and includes 10 participants with ulcers at the foot sole, who exercises for 10 weeks, twice a week, in a structured program, closely supervised by a physiotherapist. Participants´ attendance and progression in training is thoroughly recorded, as well as size and depth of ulcer.
* Participants: People with diabetes above the age of 18, resident in the Community of Copenhagen.
* Data:

Independent variables:

* Age
* Gender

Dependant variables with registration of following parameters at baseline and at end of program:

* Muscle strength measured both isometric and dynamically
* Area of ulcer
* HbA1c
* Toe pressure

Collecting data:

Data will be registrated in two phases: at phase 1(pilot study)with 10 participants, and at phase 2 (RCT study), with suitable amount of participants based on power calculations after revision of methods based on experiences from the pilot study. For all participants the program includes two attendances at inclusion and at the end of program. First examination takes place at Copenhagen University Hospital Hvidovre,and includes measuring toe pressure and level of glucoses(HbA1c). Second examination includes measuring of area of ulcer by nurse and assessment of neuropathy, muscle strength, aerobic function, and screening for performing activities in daily life by physiotherapist, at Rehabilitation Centre Vanloese. Same examinations take place at end of program.

* Intervention

Phase 1(feasibility of exercise program):

After initial examinations, 10 participants with foot ulcers participates in standardized group training for 10 weeks, for one hour, twice a week. The program consists of warming-up and aerobic exercise on stationary bike(15 min), with submaximal training at 60-70%, estimated with Borg Scale. Resistance is low to minimize weightbearing on footbed and participants will instead strive for high cadence to achieve appropriate effect from exercise. The resistance training part of the program (35 min) will include training in exercise equipment for the following muscle groups:

* flexors and extensors of knee
* abductors of hip
* extension over glenohumeral joint and upper back (low row)

In no exercise equipment is there pressure on footbed. Resistance level is 15 RM for the first three weeks and hereafter is progression up to 10RM sought.

Strengthening of ankle dorsiflexors with resistance from elastic band is also part of resistance exercises.

The last part of each exercise occasion(10 min) consists of exercises for ankle joint mobility (flexion, dorsiflexion, inversion, eversion). The prescribed ulcer treatment by nurse continues as usual.

Phase 2:

With revised manual a larger study will be implemented and by computerized block randomization, to equally sized groups with all new participants, whereas the intervention group follows the revised, standardized training program as in phase 1, besides the prescribed ulcer treatment by nurse, and the control group follows prescribed ulcer treatment and maintains usual activity level.

For phase 2 the primarily effect target is whether resistance- and aerobic training in a population of people with diabetes with foot ulcers shows effect on muscle strength, aerobic function and balance.

The statistical analysis will be repeated measures variance analysis (ANOVA) for determining effect of resistance- and aerobic training as balance score between baseline and at end of program.

3.8 Data processing and analysis: Data will be collected and entered to SPSS by project manager. Statistical analysis will be repeated measures variance analysis (ANOVA) for determining effect of resistance- and aerobic training.

ELIGIBILITY:
Inclusion Criteria:

* patients with stable, diabetic ulcer on foot sole in treatment by nurse
* who speaks and understands Danish
* are able to give consent
* are allowed to walk at least short distances
* above 18 years old
* are able to participate in group exercises

Exclusion Criteria:

* patients with infection in ulcer
* with critical ischemia(<40 mm Hg toe pressure)
* not accepted to participate by answering doctor with regards to safety on renal, heart or eye function
* dyspnea to an extent, that affects speaking
* wheel chair user

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-02; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
10 Repetition Maximum (RM)for knee flexor, knee extensor, hip abductor, low row | 10 weeks after entering exercise programme
  Change in strength measured by 10 Repetition Maximum(RM)
Patient Specific Functional Scale(PSFS) | 10 weeks after entering exercise programme
  Change in ability to perform everyday life tasks, scale from 0-10, 0=can not perform, 10=same level as before ulcer
Endurance cycling on stationary bike | 10 weeks after entering exercise programme
  Change in number of km in 12 min
Number of ankle dorsiflexion repetitions | 10 weeks after entering exercise programme
  Change in maximum number of repetitions with elastic band
Ulcer area | 10 weeks after entering exercise programme
  Change in ulcer area measured in cm2

SECONDARY OUTCOMES:
Participant satisfaction measured by Numeric Rating Scale(NRS) | 10 weeks after entering exercise programme
  Participant scores satisfaction with programme 0=lowest possible satisfaction 10=highest possible satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Kajsa Lindberg, PT, Principal Investigator — Vanloese Rehabilitation Centre, Community of Copenhagen; Morten Tange Kristensen, ph d, senior researcher, Study Chair — Dpt of Physiotherapy and Dpt of Orthopaedic Surgery, University Hospital of Copenhagen, Capital Region of denmark
Locations (1):
- Rehabilitation Centre Vanloese, Copenhagen, Vanloese, Denmark